CLINICAL TRIAL: NCT02438631
Title: Placental Passage and Disposition of Drugs: A Physiology-based Approach
Acronym: PIANO
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Janssen Pharmaceuticals (Industry); Merck Sharp & Dohme LLC (Industry); PENTA Foundation (Network); Top sector Life Sciences & Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: PIANO
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Pregnancy
Keywords: placenta; placental passage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Placental tissue is retained, limited sample. DNA will not be analysed.
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators aim to integrate the outcomes in physiology-based pharmacokinetic (PBPK) models to put the generated data into context with medical conditions that require maternal or fetal drug therapy (e.g. HIV). These models will be validated with available 'real-life' maternal and fetal PK data, such as data from the PANNA network.

PBPK models of drug therapy during pregnancy will provide a powerful tool to 1.) assist in designing rational dosing adjustments, 2.) prevent intervention-based research in pregnant women in the future, and 3.) guide future development of new molecular entities (e.g. preventing heavy investment in drugs with high predicted fetal exposure and potentially toxic effects in utero).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age > 18
* Signed informed consent
* >38 weeks pregnant

Exclusion Criteria:

* Retained placenta
* HIV infected
* Known hepatitis C infection
* Multiple pregnancy
* Congenital birth defects child
* Sectio EXIT procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
placental transfer | at delivery
  1.) An ex-vivo placenta perfusion model will be used to estimate placental passage of drugs
histological profiling | at delivery
  Histological and protein profiling experiments will be conducted to investigate factors that may influence the placental passage and disposition of drugs (e.g. the abundance, localization and inter-individual variation of expression of enzymes and transporters).
in vitro experiments | at delivery
  Furthermore, in vitro experiments will be conducted to estimate the pharmacodynamic effects of drugs on the placental barrier function itself (e.g. whether exposure to drugs can induce/reduce the expression of enzymes and transporters, as has been reported for several organs, such as the liver, intestine and kidney).

CONTACTS AND LOCATIONS:
Overall Officials: J van Drongelen, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands